CLINICAL TRIAL: NCT04286854
Title: Echocardiographic Assessment of the Right Ventricle in Healthy Subjects During Stress Test in the Mexican Population
Acronym: ECORVStressMx
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Miguel Ayala León (Network)
Collaborators: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Sponsor-Investigator, Miguel Ayala León, cardiovascular critical care unit director, Hospital Beneficencia Espanola de Puebla
Organization: Hospital Beneficencia Espanola de Puebla (Network)
Other Study IDs: Cardiologia-001
Record Dates: First submitted 2020-02-24; First posted 2020-02-27 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Echocardiography, Stress; Reference Values
Keywords: Echocardiography, Stress; Right ventricle; Mexican population
MeSH Terms: interventions — Echocardiography, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Stress echocardiography with semi-supine bicycle — The patient is accelerating against a workload that gradually increases at a constant rate, during the exercise the images will be obtained by echocardiography.
  The patient begins with 25 Watts with increments of 25 Watts every 3 minutes, continuing the exercise until significant electrocardiographic changes occur or the patient starts with symptoms.

SUMMARY:
The echocardiographic indices of the right ventricle function vary significantly with demographic and anthropometric of each population factors and are associated with poor prognosis in several cardiovascular diseases.

This study aims to investigate exercise-induced changes in echocardiographic indices of the right ventricle function in healthy volunteers and establish the reference values to the Mexican population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women
* Age ≥18 years and < 45.
* No history or symptoms of cardiovascular or lung disease
* No cardiovascular risk factors, that is, arterial systemic hypertension, smoking, diabetes, dyslipidemia
* No ongoing or previous cardio or vasoactive treatment
* Normal ECG
* Normal physical examination
* Able to use the semi-supine exercise bicycle
* Able to give informed consent

Exclusion Criteria:

* Tricuspid regurgitation more than mild
* Poor acoustic window.
* Professional sports activity
* Pregnancy
* Obesity (body mass index [BMI], ≥30 kg/m2).
* No knowledge of serum lipid or glucose levels at any time
* Inability to provide consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: -The sample will be selected from a group of volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Response of diastolic and systolic function of the right ventricle during stress test by echocardiography in a healthy Mexican Cohort | 1 hour
  The following variants will be measured by echocardiography during rest and peak exercise
  Left atrium (LA)
  * LA volume index Left ventricle (LV)
  * LV telediastolic diameter
  * LV telesystolic diameter
  * LV posterior wall Right atrium (RA)
  * RA area Right ventricle (RV)
  * RV basal dimensión
  * RV mid cavity dimension;
  * RV longitudinal dimension
  * Distal, RV outflow tract dimension at the distal or pulmonic valve level
  * Proximal RV outflow tract dimension at the proximal subvalvular level
  * Tricuspid annular plane systolic excursion
  * RV free Wall strain
  * Inferior cava vein PW Doppler
  * E wave mitral
  * A wave mitral
  * E wave /A wave mitral
  * E-wave at mitral annulus (cm/s)
  * E-wave at mitral annulus / A-wave at the mitral annulus
  * E wave/ E-wave at the mitral annulus
  * E tricuspid (E)
  * A tricuspid (A)
  * E/A
  * E-wave at the tricuspid annulus
  * Systolic pulmonary artery pressure
  * Mean pulmonary artery pressure
  * Stroke volume
  * Cardiac output

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Beneficencia Española de Puebla, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No